CLINICAL TRIAL: NCT06642948
Title: Evaluating the Efficacy of Structured Exercise Interventions in Alleviating Aromatase Inhibitor-Induced Arthralgia in Breast Cancer Survivors: A Randomized Controlled Trial
Brief Title: AI-based Skeleton Recognition System for Rehabilitation Exercise in Breast Cancer Survivors: A Randomized Controlled Trial
Acronym: AiRE-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiang Lingyun, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13825489001123; 82272922 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Musculoskeletal Symptoms; Breast Cancer; Endocrine Therapy; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Patients in the intervention group will engage in a home-based exercise program in addition to standard rehabilitation guidance.
  Interventions: Other: Motor rehabilitation based on ai visual recognition
- Control group (No Intervention): Patients will receive guidance on breast cancer endocrine therapy-related knowledge, including exercise rehabilitation for bone and joint symptoms (including the freedom to choose the form, type, and intensity of exercise), psychological counseling, and health education.

INTERVENTIONS:
Other: Motor rehabilitation based on ai visual recognition — Patients in the intervention group will engage in a home-based exercise program in addition to standard rehabilitation guidance. Initially, patients will be provided with exercise materials developed by the intervention team, one-on-one guidance via the AI rehabilitation platform, and a detailed explanation of the exercise intervention program (including its components, foundational knowledge, and benefits).The aerobic warm-up routine includes activities such as marching in place, full-body stretches, jumping jacks, side steps with arm circles, and squats with alternating punches. For the elderly, the warm-up routine is similar but also incorporates chest expansion exercises, abduction exercises, overhead reaches, lateral movements, hip extension exercises, calf raises, and additional full-body stretches.Functional training should be done 3 to 5 times per week at an intensity of RPE 3 to 4, with each session lasting 15 to 30 minutes.
  Other Names: ai visual recognition technology; exercise
  Arms: Exercise group

SUMMARY:
This study aims to develop and evaluate an artificial intelligence (AI)-based skeletal recognition system designed to support real-time, interactive rehabilitation exercise (RE programs. The goal is to mitigate musculoskeletal symptoms associated with endocrine therapy in breast cancer survivors.Endocrine therapy remains a cornerstone in the treatment of hormone receptor-positive breast cancer, typically extending over 5 to 10 years. While the therapeutic benefits of endocrine therapy are well established, agents such as aromatase inhibitors frequently induce musculoskeletal symptoms (MS), including joint pain, stiffness (particularly morning stiffness), carpal tunnel syndrome, tenosynovitis, myalgia, and muscle weakness. These symptoms, which may be continuous or intermittent, can affect both central (spine, hips, shoulders) and peripheral joints (elbows, wrists, knees, feet), severely compromising patients' quality of life (QoL). Although physical exercise has been demonstrated to alleviate these symptoms, adherence to adequate exercise regimens remains suboptimal among patients. Furthermore, there is no consensus on the optimal type, duration, or intensity of exercise interventions, and standardized protocols are lacking. Recognizing exercise as a long-term behavior, we are developing a home-based, AI-assisted rehabilitation program tailored to the specific needs of patients undergoing endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed hormone receptor-positive breast cancer (stage I, II, III).

  2. Initiation of treatment with aromatase inhibitors (e.g., anastrozole, letrozole, exemestane).

  3. Postmenopausal women, including those with surgically induced menopause. 4. Clear consciousness, no cognitive or communication impairments, and able to comply with the intervention.

  5. Informed consent obtained, with voluntary participation in the study. 6. Bone and joint symptoms with a Brief Pain Inventory (BPI) score of ≥3, or presence of at least one of the following risk factors: elevated bone turnover markers, reduced vitamin D levels, increased inflammatory cytokines, elevated C-reactive protein, or elevated rheumatoid factor.

  7. Not participating in any physical therapy or exercise-based interventions that may interfere with this study.

Exclusion Criteria:

- 1. Recurrence of breast cancer or distant metastasis. 2. Presence of other malignancies. 3. Diagnosed rheumatoid arthritis, bone and joint trauma, or other severe bone and joint diseases.

4. Bone mineral density T-score <-2.5. 5. Presence of absolute contraindications to exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 80 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Grip strength | From enrollment to the end of treatment at 12 weeks
M-SACRAH | From enrollment to the end of treatment at 12 weeks
  score for assessment and quantification of chronic rheumatic affections of the hands
WOMAC | From enrollment to the end of treatment at 12 weeks
  Western Ontario and McMaster Osteoarthritis Index
ROM | From enrollment to the end of treatment at 12 weeks
  range of motion

SECONDARY OUTCOMES:
BCTQ | From enrollment to the end of treatment at 12 weeks
  Boston Carpal Tunnel Syndrome Questionnaire
CRP | Baseline and 3 months
rheumatoid factor | Baseline and 3 months
25-hydroxyvitamin D | Baseline and 3 months
IL-1、INF-a、IL-6、IFN-a、IFN-Y | Baseline and 3 months
Bone mineral density | baseline
OPG/RANKLE SNP | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.